CLINICAL TRIAL: NCT01656668
Title: A Multicentre, Double-Blind, Placebo-Controlled, Adaptive Pivotal Study of the Efficacy and Safety of Oral BC1036 in the Management of Cough
Brief Title: Study of the Safety and Effectiveness of BC1036 Capsules to Treat Frequent Long-Term Cough
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Respicopea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC1036-001
Record Dates: First submitted 2012-07-27; First posted 2012-08-03 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Cough
Keywords: Chronic; Acute; Persistent; Longterm; Cough
MeSH Terms: conditions — Cough; Bronchiolitis Obliterans Syndrome | interventions — Theobromine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BC1036 (Experimental): BC1036 300 mg capsule capsule by mouth, twice daily, for 14 days.
  Interventions: Drug: BC1036
- Sugar Pill (Placebo Comparator): Sugar placebo capsule by mouth, twice daily, for 14 days.

INTERVENTIONS:
Drug: BC1036
  Other Names: Theobromine; CAS number 83-67-0; EV Substance code SUB15511MIG
  Arms: BC1036

SUMMARY:
The purpose of this study is to investigate the effect of BC1036 (theobromine) on cough-related quality of life and cough severity following 2 weeks' treatment.

DETAILED DESCRIPTION:
Cough is a common and disabling symptom. At any one time 20% of the population have a troublesome cough and sufferers consume 75 million doses of over-the-counter anti-tussive (anti-cough) medication annually. Chronic cough can be the presenting symptom of almost all respiratory conditions; it can also occur in the absence of overt lung pathology. The only study to grade cough severity found 7% of a general population had cough sufficient to interfere with activities of daily living on at least a weekly basis in the UK. Cross sectional studies have consistently shown that chronic cough is particularly prevalent in middle aged females.

The investigational medicinal product BC1036 (theobromine) is being developed as a non-codeine, non-narcotic treatment for persistent cough. Theobromine is a well characterised molecule with a long history of safe use both as a medicine and as a food product. As a member of the xanthine family, it bears structural and pharmacological similarity to caffeine and theophylline, both of which have long been approved for medicinal use.

This is a placebo-controlled, double-blind, parallel group study of BC1036 in subjects with persistent cough (chronic or sub-acute), treatment resistant after a routine clinical assessment as outlined in the BTS Recommendations for the Management of Cough in Adults and despite adequate treatment of any associated potential aggravating factors or without the continuance of any obvious precipitating factors. The objective is to investigate the effect of BC1036 on cough-related quality of life and cough severity following 2 weeks' treatment. It is planned to recruit 288 evaluable subjects from cough clinics, secondary and primary care centres in the UK. Subjects will receive either BC1036 or placebo over a period of 14 days.

Eligible subjects will be required to attend the clinic on five occasions: screening, baseline, days 7, 14, and a follow up visit at day 28. At every visit the subjects will complete the Leicester Cough Questionnaire (LCQ), and a cough Visual Analogue Score (VAS). Spirometry will be performed for measurement of lung function. Blood samples will be drawn for safety clinical laboratory parameters and physical examinations and ECG will be performed. Subjects should be seen for all visits on the designated day ± 1 day, except Day 28 ± 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years.
* Confirmed diagnosis of a persistent cough.
* Leicester Cough Questionnaire score of ≤ 17 at baseline.
* FEV ≥ 70% of predicted normal, at screening. See protocol Appendix 4 for formula for calculating predicted values.
* Willing to use effective contraception for the duration of the study. Female subjects who are neither surgically sterilized nor post-menopausal (defined as no menses for one year or an FSH value > 40 mIU/L) will be required to use two methods throughout the study and for 30 days after. Besides abstinence the following contraceptive methods are acceptable: hormonal (e.g. oral, injection, transdermal patch, implant, cervical ring), barrier (e.g. condom or diaphragm with spermicidal agent) or intrauterine device. If hormonal contraceptives are used they must be used from 6 weeks before the first administration of test product. Male subjects must agree to use condoms for the duration of the study and for 30 days after.
* Willing and able to give informed consent and of complying with the trial assessments and any other trial procedures.

Exclusion Criteria:

* Pregnant or lactating females.
* Major surgery within the 30 days preceding the screening visit.
* Any serious infections within the 30 days prior to the screening visit.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes, renal or hepatic disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Known hepatitis B or C or human immunodeficiency virus (HIV) or syphilis seropositivity.
* A history of serious adverse allergic reaction to any medication.
* Treatment with another investigational medicinal product within the 30 days prior to enrollment.
* Treatment with:

  * Systemic oral steroids within 7 days prior to randomisation at Visit 2.
  * Theophylline and theophylline-like agents within 7 days prior to randomisation.
  * Opiates or opioids e.g. codeine, dextromethorphan, within 7 days prior to randomisation.
  * ACE inhibitors within one month prior to the screening visit.
* Depot injection of corticosteroids within 6 weeks of the screening visit.
* History suggestive of febrile illness within the last 7 days prior to the screening visit.
* Subjects with significant sputum production (defined as more than 5 ml (~one teaspoon)/day on any three days in the screening period).
* Current smokers or past smokers who have a smoking history of > 20 pack years or stopped smoking ≤ 12 months prior to screening.
* Any pulmonary co-morbidity such as COPD, recurrent lower respiratory tract infections (≥ 2 in the 12 months prior to screening) and bronchiectasis where cough suppression may lead to sputum retention and infection.
* Any pulmonary abnormality on chest X-ray or CT scan performed in the twelve months prior to enrolment indicative of COPD, bronchiectasis etc.
* Subjects diagnosed with asthma who have suffered an exacerbation requiring hospitalisation within 4 weeks prior to screening.
* A history of cancer within the previous five years (excluding carcinoma in situ or nonmelanoma skin cancer treated by surgical excision).
* Uncontrolled hypertension (resting systolic BP > 170mmHg or resting diastolic BP > 95 mm Hg).
* A corrected QT interval of > 470ms for female subjects or of > 450ms for male subjects, calculated using the QTcF correction formula, or second degree or higher heart block on an ECG recording, at screening.
* Subjects known to have a sensitivity to methylxanthines and related compounds, or known to have exhibited an allergic response or sensitivity to cocoa-based products.
* History or presence of alcohol or substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire (LCQ) | Day 14
  Cough-related quality of life assessed using the Leicester Cough Questionnaire (LCQ). The baseline-adjusted total LCQ score at Day 14 will be used as the primary endpoint.

SECONDARY OUTCOMES:
Adapted 7-day Leicester Cough Questionnaire (LCQ) | Day 7
  Adapted 7-day LCQ to measure quality of life over the previous 7 days.
Leicester Cough Questionnaire (LCQ) | Day 28
  LCQ at Day 28 will measure quality of life over the previous 14 days.
Cough visual analogue scale (VAS) | From screening to Day 28
  VAS scores on a 100 mm scale fixed at both ends by 'no cough' and 'worst cough ever'. Assessment made at every visit.
Airway sensitivity using capsaicin challenge | Day 0 and Day 14
  Subgroup of approximately 100 subjects will be challenged with capsaicin at Day 0 and Day 14.

OTHER OUTCOMES:
Pulmonary function tests | From screening to day 28
  Pulmonary function will be measured at all visits using a calibrated spirometer. This includes Forced Expiratory Volume (FEV), Forced Vital Capacity (FVC) and peak flow.

CONTACTS AND LOCATIONS:
Overall Officials: Alyn Morice, BA(Hons) MB.B.Chir MA FRCP, Principal Investigator — Castle Hill Hospital; Fan Chung, MB, BS, MD, FRCP, DSc (PI), Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Warwick Coulson, BSc, MBBS, DipRCOG, MRCGP, Principal Investigator — Albany House Medical Centre; Alun George, MA MBBS, DRCOG, DCH, MRCGP, Principal Investigator — Staploe Medical Centre; Bernard Higgins, MB ChB, MRCP, MD, Principal Investigator — Freeman Health System; Alan Jackson, MB, BS, Principal Investigator — Sheepcot Medical Centre; Philip Marazzi, MB, BS, Principal Investigator — The Medical Centre; Ian Pavord, MB BS, MRCP, FRCP, DM, Principal Investigator — Glenfield Hospital; Surinder Birring, BSc,MBChB(Hons),MRCP,MD(PI), Principal Investigator — King's College Hospital NHS Trust; Lorcan McGarvey, MBBCh,BAOHons,MRCP,MD,CCST(PI), Principal Investigator — The Queen's University of Belfast; Richard Oliver, MB ChB, MRCGP, Principal Investigator — Ecclesfield Group Practice; Chris Strang, MB BS, D. Obst, RCOG M, Principal Investigator — Mortimer Surgery; Damien McNally, MB,BCh,BAO,DRCOG,DMH,MRCGP, Principal Investigator — Ormeau Road Health Centre
Locations (13):
- United Kingdom (13):
  - Ormeau Road Health Centre, Belfast
  - The Queen's University of Belfast, Belfast
  - Castle Hill Hospital, Cottingham
  - The Medical Centre, East Horsely
  - Sheepcot Medical Centre, Garston, Watford
  - Glenfield Hospital, Leicester
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - Mortimer Surgery, Mortimer
  - Freeman Hospital, Newcastle upon Tyne
  - Ecclesfield Group Practice, Sheffield
  - Staploe Medical Centre, Soham, Ely
  - Albany House Medical Centre, Wellingborough, Northampton

REFERENCES:
- [Derived] Morice AH, McGarvey L, Pavord ID, Higgins B, Chung KF, Birring SS. Theobromine for the treatment of persistent cough: a randomised, multicentre, double-blind, placebo-controlled clinical trial. J Thorac Dis. 2017 Jul;9(7):1864-1872. doi: 10.21037/jtd.2017.06.18. PMID 28839984